CLINICAL TRIAL: NCT06910306
Title: A Study to Assess the Feasibility and Safety of Intratumoral Diffusing Alpha Emitters for the Treatment of Recurrent Glioblastoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-GBM-01
Record Dates: First submitted 2024-09-23; First posted 2025-04-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Glioblastoma; Recurrent Gliomas
Keywords: Recurrent Glioblastoma; Brachytherapy; GBM; Alpha DaRT sources; Intratumoral Diffusing Alpha Emitters
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Intervention Model Description: This is a prospective , Multicenter , Open label, Single arm with DaRT for the treatment of Recurrent Glioblstoma .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental: DaRT seeds (Experimental): DaRT sources are inserted into the tumor according to a pre determined plan. The delivery of the DaRT Sources into the tumor is done by using a designated Alpha DaRT Applicator .
  Interventions: Device: Device :DaRT seeds

INTERVENTIONS:
Device: Device :DaRT seeds — The sources are impregnated with a layer containing Ra-224 which is well fixated to the surface of the source. Ra-224 undergoes a series of decay events with each daughter product producing an alpha particle

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for the treatment of recurrent Glioblastoma

DETAILED DESCRIPTION:
This is a Prospective Open label Single arm Multi-center interventional study. The study is designed to evaluate the Feasibility and Safety of DaRT seeds for the treatment of recurrent Glioblastoma.

A total of 10 subjects will be enrolled.

Eligible patients who meet inclusion/exclusion criteria (as assessed during the screening period) will be invited to the site for the procedure of DaRT seeds insertion and will return for a follow up visit every 2 months (+/- 7 days ) up to 12 months (4 ,6 , 8, 10 and 12 ). Survival F.U (after visit 11) will be done via phone calls every 2-3 months until (1) the start of new anti-cancer treatment, (2) disease progression or (3) death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 18 and ≤ 85 years of age
* Patients must have histologically confirmed diagnosis of WHO grade IV glioblastoma (including variants such as gliosarcoma, giant cell glioblastoma).
* Single, gadolinium-enhancing tumor recurrence ≤ 3cm in maximum diameter
* Patient not amenable for surgical resection due to any of the following but not limited reasons: patient refusal, medically ineligible, surgically too high risk due to tumor location in a deep and/or eloquent location.
* Prior history of central nervous system (CNS) radiation (standard dose) with 50.4-60 Gy delivered in 1.8 Gy-2.0 Gy fractions with concurrent temozolomide (if the patient has received a non-standard fractionation or radiation dose, such as 40 Gy in 15 fractions.
* Patients must have a time interval ≥4 months between completion of prior radiation and trial registration and have tumor progression per RANO criteria
* Patients must have a measurable disease per RANO criteria
* Estimated life expectancy is more than 6 months
* Target lesion amenable for coverage by the DaRT sources
* Patient must either have had recent subtotal surgery/biopsy following tumor recurrence (at least 6 weeks from trial registration) or must have shown unequivocal radiographic evidence for tumor progression by contrast-enhanced MRI scan within 21 days prior to trial registration. If surgery was performed, must have a post-operative MRI scan within 21 days prior to trial registration.
* Patients have recovered from prior therapy side effects and must be at least 4 weeks post administration of chemotherapies or investigational agents with the exception of nitrosureas (such as Carmustine, Fotemustine, Lomustine) which requires 42 days of washout.
* Karnofsky performance score (KPS) of at least 60 documented within 14 days prior to trial registration
* Patients must have adequate biological parameters as demonstrated by the following blood counts at initial screening obtained ≤ 14 days prior to starting treatment Absolute neutrophil count (ANC) ≥ 1.5 × 109/L Platelet count ≥ 100,000/mm3 (80 × 109/L) Hemoglobin (Hgb) ≥ 9 g/dL.
* Patients must have the following blood chemistry levels at initial screening obtained ≤ 14 days prior to starting treatment AST (SGOT), ALT (SGPT) ≤ 2.5 × upper limit of normal range (ULN) Total bilirubin ≤ 1.5 × ULN
* Effective contraception must be used by both male and female patients while on the study and for up to 3 months following treatment
* Patient must have been informed about the nature of the study, and must have agreed to participate in the study, and signed the Informed Consent Form (ICF) prior to participation in any study-related activities

Exclusion Criteria:

* Medical contraindication to MRI (cardiac devices are allowed if MRI compatible)
* More than 3 relapses per RANO criteria
* Acquired and or genetic clinical bleeding tendency
* Suspicious of infratentorial or leptomeningeal or intraventricular disease
* Concomitant chemotherapy or any other systemic therapy not allowed in the protocol
* Recent or current (within 6 weeks) therapy with VEF or a VEGFR inhibitor
* Immunocompromised state due to either transplant or AIDS
* Prior allergic reaction to the study drugs
* History of hypertensive crisis or hypertensive encephalopathy
* Uncontrolled hypertension (defined as either >150 mm/Hg for systolic and >90mm/Hg for diastolic)
* History of a non-healing wound, ulcer, gastrointestinal bleed (> grade 3), traumatic injury, or bone fracture within 90 days prior to registration Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT
* High probability of protocol non-compliance (in opinion of investigator)
* Pregnancy or lactation
* Collagenous diseases, specifically systemic lupus erythematosus, scleroderma, or dermatomyositis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility - DaRT seed placement | From day 0 until 12 months
  Feasibility will be determined according to the rate of successful placement of Alpha DaRT sources into brain tumors.
Safety - Adverse events | From day 0 until 12 months
  Safety will be determined according to incidence of acute grade 3 or greater unanticipated Adverse Events (AE) according to CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Toxicity profile | within 4 weeks of completion of postoperative radiotherapy
  according to CTCAE v5.0
Radiographic local tumor control | from 1 month following surgery and onwards
  per RANO criteria
Rate of pseudo-progression at first post-implant scan | 1 month following surgery
  RANO criteria
Overall survival | up to 12 months post implant

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States